CLINICAL TRIAL: NCT05956847
Title: The Role of Extracellular DNA (ecDNA) in the Occurrence and Development of Gastric Cancer: an Exploratory Multicenter Prospective Observational Clinical Study
Brief Title: The Role of Extracellular DNA (ecDNA) in the Occurrence and Development of Gastric
Status: Recruiting | Type: Observational
Sponsor: Xijing Hospital (Other)
Collaborators: Yuncheng Central Hospital (Other); Xi'an Honghui Hospital (Other); Xi'an No.9 Hospital (Unknown); Xi'an No.3 Hospital (Other Government); Xijing 986 Hospital (Unknown)
Responsible Party: Sponsor
Other Study IDs: Gang Ji -3
Record Dates: First submitted 2023-07-07; First posted 2023-07-21 (Actual); Last update posted 2023-08-29 (Actual); Status verified 2023-06

CONDITIONS: Gastric Cancer; Precancerous Lesion of Digestive Tract; Extrachromosomal DNA
MeSH Terms: conditions — Stomach Neoplasms | interventions — Gastroscopy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 5 Years
Biospecimen Retention: Samples With DNA — Gastroscopy biopsy specimen，venous blood，gastric cancer tissue
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Gastric precancerous lesions，Normal gastric mucosal tissue and gastric cancer tissues: Normal gastric mucosal tissue Gastric precancerous lesions:Atrophic gastritis, non Atrophic gastritis, intestinal metaplasia, dysplasia gastric cancer tissues
  Interventions: Procedure: gastroscopy

INTERVENTIONS:
Procedure: gastroscopy — When performing gastroscopy, the endoscopist will perform a biopsy based on the condition of gastric mucosal lesions, with one specimen retained and the remaining specimens subjected to pathological examination
  Other Names: Pathological biopsy

SUMMARY:
ECDNA is almost non-existent in normal cells, but exists in nearly half of human cancer cells, indicating that studying such abnormal DNA is of great significance for our understanding of tumor formation and evolution. The changes in ecDNA expression in intestinal type gastric cancer may be closely related to the occurrence and development of gastric cancer. Dynamic monitoring of changes in ecDNA expression in the gastric mucosa may help predict the occurrence of gastric cancer and guide subsequent treatment. By collaborating with multiple endoscopic centers to conduct gastroscopy biopsies on patients with gastric precancerous lesions, we aim to further explore the role of ecDNA in the occurrence and development of gastric cancer through continuous follow-up.

ELIGIBILITY:
Inclusion Criteria:

1. Age: 18-80 years old;
2. Patients who plan to undergo gastroscopy at the endoscopic center and patients who undergo surgical treatment for gastric adenocarcinoma;
3. Endoscopy doctors believe that pathological biopsy is necessary to clarify the pathological diagnosis;
4. No serious diseases or other systemic malignancies in terms of physical and mental health;
5. More than one item of non Atrophic gastritis, Atrophic gastritis, intestinal metaplasia, heterogeneous hyperplasia (low grade intraepithelial neoplasia and high grade intraepithelial neoplasia), and gastric adenocarcinoma;
6. Sign an informed consent form;

Exclusion Criteria：

1. Pathological results indicate other malignant tumors of the stomach, such as stromal tumors and lymphoma;
2. The patient and their family members do not agree to use the specimen for later research projects;
3. Before gastroscopy or surgery, neoadjuvant therapy or combined with other malignant tumors;
4. Non R0 resected gastric cancer patients;
5. Pregnant or lactating women;
6. Have a history of drug abuse such as alcohol and tobacco.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The population included in this study is mainly healthy patients who underwent gastroscopy at endoscopic centers, some of whom may develop gastric cancer during follow-up. At the same time, we will collect mucosal samples from volunteers who underwent gastroscopy but had normal gastric mucosa, and we will also collect gastric cancer tissue samples after surgical resection in our department
Sampling Method: Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2023-08-10 (Actual); Primary Completion 2028-07-20 (Estimated); Study Completion 2030-07-30 (Estimated)

PRIMARY OUTCOMES:
Changes in ecDNA content in different gastric precancerous lesions | 2023/11-2024/11
  Compare the differences in ecDNA in gastric mucosal tissue at different stages of gastric precancerous lesions, and explore the role of ecDNA in disease progression after 5 years of follow-up

CONTACTS AND LOCATIONS:
Overall Officials: Guo Xin, Principal Investigator — Xijing 986 Hospital; Wang Tongfei, Principal Investigator — Xi'an No.3 Hospital; Hao Junfeng, Principal Investigator — Xi'an No.9 Hospital; Shi Yupeng, Principal Investigator — Xi'an Honghui Hospital; Gao Xiaopeng, Principal Investigator — Yuncheng Central Hospital
Locations (1):
- Xijing Hospital of Digestive Diseases, Xi'an, Shaanxi, China

IPD SHARING:
Plan to Share IPD: Undecided